CLINICAL TRIAL: NCT05000606
Title: The Effect of a Home Visit Program for Caregivers of Asthmatic Patients on Perceived Care Burden
Brief Title: A Home Visit Program and Perceived Care Burden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ayaz Alkaya, Professor, Faculty of Nursing, Nursing Department, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 77082166-604.01.0
Record Dates: First submitted 2021-07-29; First posted 2021-08-11 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2021-08

CONDITIONS: Burden
Keywords: asthma; burden; caregiver; education; home visit
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A home visit program (Experimental): A home visit program including five visits over three months were performed.
  Interventions: Other: A home visit program
- Control (No Intervention): No other intervention was applied to the control group other than the standard education given in the outpatient clinic

INTERVENTIONS:
Other: A home visit program — A home visit program including education and counseling was applied. A total of five home visits over three months were performed.
  Arms: A home visit program

SUMMARY:
The aim of this study was to determine the effect of a home visit program provided to the caregivers of asthmatic patients on the perceived care burden. A randomized controlled trial was used. The sample consisted of 30 participants in the intervention group and 30 participants in the control group. A home visit program including education and counseling was applied to participants in the intervention group.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of a home visit program provided to the caregivers of asthmatic patients on the perceived care burden. A randomized controlled trial was used. The sample consisted of 30 participants in the intervention group and 30 participants in the control group. A home visit program including education and counseling was applied to participants in the intervention group. A total of five home visits over three months were performed. Data were collected by a personal information form, and the Zarit Caregiver Burden Scale (ZCBS).

ELIGIBILITY:
Inclusion Criteria:

* giving care to a patient who was poorly controlled or uncontrolled asthma
* giving care to a patient who used an inhaler
* age 18 or over
* volunteering to participate to the study

Exclusion Criteria:

* having a disease with a neuro-psychiatric diagnosis
* having vision and hearing problems

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Zarit Caregiver Burden Scale | Baseline
  The scale consists of 18 questions. The minimum test score is 0 and the maximum score is 72. Care burden increases as the score from the scale increases.
Zarit Caregiver Burden Scale | Change from Baseline Perceived Care Burden Scores at 1 month
  The scale consists of 18 questions. The minimum test score is 0 and the maximum score is 72. Care burden increases as the score from the scale increases.
Zarit Caregiver Burden Scale | Change from 1 month Perceived Care Burden Scores at 3rd months
  The scale consists of 18 questions. The minimum test score is 0 and the maximum score is 72. Care burden increases as the score from the scale increases.

IPD SHARING:
Plan to Share IPD: No